CLINICAL TRIAL: NCT03842917
Title: SAlt Diet and Various Biomarkers Effects on Blood Pressure and Proteinuria During Inhibition of VEGF)
Acronym: SAVE
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18/SAVE; 2018-A03137-48 (Other: IdRCB)
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Patient Starting Bevacizumab; Cancer
Keywords: Cancer; bevacizumab; blood pressure; proteinuria
MeSH Terms: conditions — Neoplasms; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and blood samples will be drawn to measure proteinuria and concentration of various biomarkers (as listed above)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient starting bevacizumab treatment for cancer: Taken biological samples (urine and blood) and blood pressure measurement on patients starting bevacizumab treatment for cancer
  Interventions: Other: Biological samples; Other: Blood pressure measurement

INTERVENTIONS:
Other: Biological samples — Urine and blood samples
Other: Blood pressure measurement — Home blood pressure self-measurement and hospital blood pressure measurement

SUMMARY:
Bevacizumab is an anti-angiogenic treatment used to treat various solid cancers. Previous studies have shown that this treatment may have adverse effects like hypertension and proteinuria.

This is an exploratory study aiming to better understand the relationship between various biomarkers and blood pressure changes and proteinuria measured for 4 to 6 weeks after the first infusion of anti-VEGF therapy with bevacizumab.

DETAILED DESCRIPTION:
Participants will be invited to participate to this research study by their oncologist within 1 to 2 weeks before starting bevacizumab treatment, as part of standard treatment. They will finish the research at the end of the third infusion of bevacizumab.

Patients will perform a home blood pressure self-measurement over three days and will collect urine over 24 hours prior to the start of each bevacizumab infusion at cycles 1, 2 and 3. Blood pressure measurements will also be performed during each bevacizumab infusion and blood tests will be performed before each infusion to measure the following biomarkers:

* Salt consumption as estimated by 24-hour natriuresis measured before each of the first 3 infusions
* 24 hours aldosterone excretion measured before the first and third infusions
* plasma methoxylated derivatives measured before the first and third infusions
* NTproBNP measured before the first and third infusions
* 24 hours urinary free cortisol measured before the first and third infusions
* bevacizumab trough concentration measured before the first three bevacizumab infusion

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* With a solid cancer for which a treatment with bevacizumab (Avastin®) is indicated in accordance with its marketing authorization

Exclusion Criteria:

* Renal cancer
* Recent changes in antihypertensive treatment(s) in the last month, with the exception for diuretics where treatment stability of at least 3 months will be required
* Patients who do not wish to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid cancers who will be starting treatment with bevacizumab as part of the standard treatment
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Home blood pressure measurement | before the initiation of bevacizumab and before each bevacizumab infusion, up to 10 weeks
  Home blood pressure (systolic, diastolic) before each bevacizumab infusion, as the mean of 3 measures in the morning and 3 measures in the evening, over 3 days

SECONDARY OUTCOMES:
in-hospital blood pressure measurement | before the initiation of bevacizumab and before each bevacizumab infusion, up to 10 weeks
  Standardized measurement of in-hospital blood pressure (systolic, diastolic) and heart rate during bevacizumab infusion
24-hour proteinuria | before the initiation of bevacizumab and before each bevacizumab infusion, up to 10 weeks
  Measurement of 24 hours proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Theodora BEJAN-ANGOULVANT, MD-PhD, Study Director — University Hospital, Tours
Locations (3):
- France (3):
  - Medical Oncology Service, University Hospital, Tours, Tours
  - Oncological Gastroenterology Service, University Hospital, Tours, Tours
  - Pneumology, University Hospital, Tours, Tours